CLINICAL TRIAL: NCT03811665
Title: A Prospective Randomized Pilot Trial of Stereotactive Body Radiation Therapy Versus Radiofrequency Ablation for the Management of Small Renal Masses.
Brief Title: Stereotactic Body Radiation Therapy Versus Radiofrequency Ablation for Small Renal Masses
Acronym: SBRT vs RFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Principal Investigator, Anil Kapoor, Principal Investigator, St. Joseph's Healthcare Hamilton
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RADSTER
Record Dates: First submitted 2018-11-13; First posted 2019-01-22 (Actual); Last update posted 2021-12-16 (Actual); Status verified 2021-12

CONDITIONS: Small Renal Masses (SRM)
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stereotactic body radiation therapy (SBRT) (Experimental)
  Interventions: Radiation: Stereotactive body radiation therapy
- Radiofrequency Ablation (RFA) (Active Comparator)
  Interventions: Procedure: Radiofrequency Ablation

INTERVENTIONS:
Procedure: Radiofrequency Ablation — RFA probe will create an ablation zone of a 1.0 cm diameter beyond the maximum CT-measured tumor diameter. The generator will modulate power up to 150 W in reach average ablative temperature of 105oC. Tumors will be treated for two cycles of 8 minutes duration each upon reaching target temperatures.
  Other Names: RFA
  Arms: Radiofrequency Ablation (RFA)
Radiation: Stereotactive body radiation therapy — The Gross Tumour Volume (GTV) is defined as the visible tumour seen on the planning CT simulation. No clinical target volume (CTV) for microscopic disease is necessary. The internal target volume (ITV) accounts for changes in tumour position due to respiration, and is assessed on 4DCT. The planning target volume (PTV) will be a standard 0.5 cm around the ITV.
  Other Names: SBRT
  Arms: Stereotactic body radiation therapy (SBRT)

SUMMARY:
The execution of this study is pertinent to evaluating SBRT's short- and long-term efficacy and safety in the treatment of SRMs. This study will be the first to compare RFA and SBRT in the treatment of SRMs.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age and capable of providing informed consent
* Patients scheduled for treatment of their SRM using SBRT or RFA
* Patients who received a biopsy of their SRM prior to their scheduled SBRT or RFA treatment
* Patients who are willing to have a biopsy 12 months post-procedure
* Patients with renal tumor(s) ≤ 4.0 cm

Exclusion Criteria:

* Patients with large renal tumor(s)>4.0 cm
* Patients who are unable to have a general anesthetic
* Patients who did not receive a biopsy of their SRM prior to their scheduled SBRT or RFA treatment
* Patients who are unable to comply with post-operative and/or follow-up protocol/phase of study
* Evidence of metastatic disease
* Uncorrectable bleeding diathesis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Treatment failure | 12 Months
  Failure will be defined as enhancement of ablated tissue greater than 10 Hounsfield units by CT contrast.
Overall Survival | 12 Months
  Defined as post-procedural survival.
Disease free survival | 12 Months
  Defined as disease-free survival rate after a single procedure
Disease recurrence | 12 Months
  Defined as disease recurrence rate after a single procedure, including positive biopsy result.

SECONDARY OUTCOMES:
Tumour Size | 12 Months
  Average percentage decrease in tumor size.
Renal Function -eGFR | 12 Months
  Change in eGRF measured by mL/min/1.73m2.
Renal Function - Serum Creatinine | 12 Months
  Change in serum creatinine level measured by umol/L.
Renal Function - Creatinine Clearance | 12 Months
  Change in creatinine clearance measured by ml/minute.
Complication Rate | 12 Months
  Intra and post intervention complication rates will be documented in terms of nausea, vomiting, diarrhea, hematuria, hemorrhage (requiring or not requiring transfusion), perinephric hematoma, ureteral strictures, loss of a renal unit, urinary leak, bleeding, fever and flulike symptoms, stomach/bowel ulceration, ureteropelvic junction obstruction, and upper pole hydrocalycosis.
Number of patients that experienced an adverse event. | 12 Months
  Defined by any adverse event listed in the CTCAE.
Change in score for quality of life | 12 Months
  Defined by the generic EuroQol (EQ-5D) questionnaire that is a standardized measure of health. A scale of 0-100 (0 being the worse health, and 100 being the best health), is used for a patient to define their overall health and wellbeing.
Duration of hospital stay | Days
  Duration of length of hospital stay (if applicable)
Cost analysis | 12 Months
  Defined by total cost of procedure and any associated related adverse events post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Anil Kapoor, MD FRCSC, Principal Investigator — St. Joseph's Healthcare Hamilton
Locations (1):
- McMaster Institute of Urology - St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cassim R, Bansal R, Millan B, Mironov O, Ahir P, Tajzler C, Hoogenes J, Matsumoto ED, Quan K, Kapoor A, Swaminath A. A Randomized Trial of Stereotactic Body Radiation Therapy vs Radiofrequency Ablation for the Treatment of Small Renal Masses: A Feasibility Study (RADSTER). Urology. 2025 Jun;200:118-124. doi: 10.1016/j.urology.2025.02.053. Epub 2025 Mar 7. PMID 40058468